CLINICAL TRIAL: NCT06072170
Title: Adaptive Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of Single Ascending Doses of Kratom in Healthy, Nondependent, Adult Recreational Polydrug Users With Opioid Experience
Brief Title: Single Ascending Doses of Kratom in Healthy Nondependent Adults With Opioid Experience
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Altasciences Company Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 75F40121C00199 (FDU-P4-117); 75F40121C00199 (Other: DHHS / FDA / OAGS / DAO)
Record Dates: First submitted 2023-09-19; First posted 2023-10-10 (Actual); Results first posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Safety; Pharmacokinetics; Pharmacodynamics
Keywords: Kratom; Mitragynine; Botanical substance; Single Ascending Dose
MeSH Terms: interventions — mitragynine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The treatment assignment (active or placebo) will not be known by the study participants. Study participants will be informed of the dose range they could receive but will not be informed of the actual dose assigned to them.
  Furthermore, the randomization code will not be available to the Investigator and clinical staff involved in the collection, monitoring, revision, or evaluation of AEs, as well as clinical staff who could have an impact on the outcome of the study including the pharmacokineticist (or delegate) and biostatistician, until all the case report form (CRFs) have been approved and signed and the bioanalytical phase of the study has been completed.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort 1, 1 g of Kratom (Experimental): A total of 6 subjects will receive an oral single dose administration of the active product
  Interventions: Drug: Kratom
- Cohort 2, 3 g of Kratom (Experimental): A total of 6 subjects will receive an oral single dose administration of the active product
  Interventions: Drug: Kratom
- Cohort 3, 8 g of Kratom (Experimental): A total of 6 subjects will receive an oral single dose administration of the active product
  Interventions: Drug: Kratom
- Cohort 4, 10 g of Kratom (Experimental): A total of 6 subjects will receive an oral single dose administration of the active product
  Interventions: Drug: Kratom
- Cohort 5, 12 g of Kratom (Experimental): A total of 6 subjects will receive an oral single dose administration of the active product
  Interventions: Drug: Kratom
- Placebo (Placebo Comparator): A total of 2 subjects per cohort will receive an oral single dose administration of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Kratom — Single administration thirty minutes after the start of a high-fat breakfast
  Arms: Cohort 1, 1 g of Kratom; Cohort 2, 3 g of Kratom; Cohort 3, 8 g of Kratom; Cohort 4, 10 g of Kratom; Cohort 5, 12 g of Kratom
Drug: Placebo — Single administration thirty minutes after the start of a high-fat breakfast
  Arms: Placebo

SUMMARY:
Kratom (Mitragyna speciosa) is a plant often used to self-treat conditions such as pain, coughing, diarrhea, anxiety and depression, opioid use disorder, and opioid withdrawal. Due to limited data availability, the goal of this clinical trial is to learn about safety, pharmacokinetics (what the body does to the drug) and pharmacodynamics (what the drug does to the body) of Kratom in adult recreational polydrug users with opioid experience.

DETAILED DESCRIPTION:
This is a phase I, single-dose, randomized, adaptive, double-blind, placebo-controlled, single ascending dose (SAD), sequential group study in adult recreational polydrug users with opioid experience performed at a single study center.

This study will consist of five cohorts.

Forty subjects are planned to participate. Eight subjects will participate in each cohort.

Within each cohort, 6 subjects will be randomized to receive Kratom and 2 subjects will be randomized to receive placebo. Each subject will be involved in the study for up to approximately 37 days (including screening).

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form (ICF)
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Healthy adult male or female
4. Current nondependent, polydrug recreational user who has used opioid drugs for recreational (nontherapeutic) purposes (i.e., for psychoactive effects) and has a history of recreational use of at least 2 or more of any of the perception-altering (e.g., lysergic acid diethylamide [LSD], kratom, cannabis, dronabinol, ketamine, phencyclidine [PCP], dextromethorphan, 3,4 methylenedioxymethamphetamine [MDMA], mescaline, psilocybin, tryptamine derivatives or ring-substituted amphetamines with perception altering effects) or stimulant (e.g., cocaine, amphetamine, methamphetamine, methylphenidate, methcathinone, and other synthetic cathinones) drugs
5. If male, meets one of the following criteria:

   1. Is able to procreate and agrees to use one of the accepted contraceptive regimens and not to donate sperm from study drug administration to at least 90 days after study drug administration. An acceptable method of contraception includes one of the following:

      * Abstinence from heterosexual intercourse
      * Double-barrier method (e.g., male condom with spermicide or male condom with a vaginal spermicide [gel, foam, or suppository]) Or
   2. Is unable to procreate; defined as surgically sterile (i.e., has undergone a vasectomy at least 180 days prior to study drug administration)
6. If female, meets one of the following criteria:

   1. Is of childbearing potential and agrees to use an acceptable contraceptive method. Acceptable contraceptive methods include:

      a1. Abstinence from heterosexual intercourse from the Screening visit through to at least 30 days after study drug administration

      a2. One of the following contraceptive methods, used from at least 28 days prior to the Screening visit through to at least 30 days after study drug administration:
      * Systemic contraceptives (combined birth control pills, injectable/implant/insertable hormonal birth control products, or transdermal patch)
      * Intrauterine device (with or without hormones)
      * Male partner vasectomized at least 6 months prior to the Screening visit

      a3. One of the following double-barrier contraceptive methods, used from the Screening visit through to at least 30 days study drug administration:
      * Male condom plus spermicide
      * Diaphragm plus spermicide
      * Cervical cap plus spermicide
   2. Is of non-childbearing potential, defined as surgically sterile (i.e., has undergone complete hysterectomy, bilateral oophorectomy, or tubal ligation), or is in a postmenopausal state (i.e., at least 1 year without menses without an alternative medical condition prior to the Screening visit and follicle stimulating hormone levels ≥ 40 mIU/mL at Screening)
7. Body mass index (BMI) within 18.0 kg/m2 to 34.0 kg/m2, inclusively at Screening
8. Minimum weight of 50.0 kg at Screening
9. Have no clinically significant diseases captured in the medical history or evidence of clinically significant findings on the physical examination (including vital signs, oxygen saturation [SpO2], and respiratory rate) and/or ECG, as determined by an Investigator

Exclusion Criteria:

1. Difficulty swallowing capsules
2. Female who is lactating
3. Female who is pregnant according to the pregnancy test at Screening or prior to study drug administration
4. Male with female partner who is pregnant, lactating, or planning to become pregnant during this study or within 90 days after study drug administration
5. History of significant hypersensitivity to kratom or any related products (including excipients of the formulations) as well as severe hypersensitivity reactions (like angioedema) to any drugs
6. Presence or history of significant gastrointestinal, liver or kidney disease, or surgery that may affect drug bioavailability with the exception of cholecystectomy that is permitted at the discretion of an Investigator
7. History of significant hepatic, renal, cardiovascular, pulmonary, hematologic, neurological, psychiatric, gastrointestinal, endocrine, immunologic, ophthalmologic, or dermatologic disease
8. Presence of any significant respiratory illness or presence or history of chronic respiratory disease (e.g., upper respiratory illness, sleep apnea, emphysema, asthma) at Screening (subjects with acute respiratory illness may be rescheduled upon resolution at the discretion of an Investigator)
9. History of substance or alcohol moderate to severe use disorder (excluding nicotine and caffeine) within the past 2 years, as defined by the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5)
10. Is a heavy smoker (> 20 cigarettes per day) and/or is unable to abstain from smoking or unable to abstain from the use of prohibited nicotine-containing products for at least 1 hour before and 8 hours after study drug administration (including e-cigarettes, pipes, cigars, chewing tobacco, nicotine topical patches, nicotine gum, or nicotine lozenges)
11. Regularly consumes excessive amounts of caffeine or xanthines, defined as greater than 6 servings (1 serving is approximately equivalent to 120 mg of caffeine) of coffee, tea, cola, or other caffeinated beverages per day
12. History of suicidal behavior within 2 years of Screening, showing suicidal tendency as per the C-SSRS administered at Screening, or is currently at risk of suicide in the opinion of an Investigator
13. Presence of clinically significant ECG abnormalities at the Screening visit, as defined by medical judgment. Note: QT corrected according to Fridericia's formula (QTcF) interval of > 450 msec in male subjects or > 470 msec in female subjects will be exclusionary. The ECG may be repeated once for confirmatory purposes if the initial value obtained exceeds the limits specified.
14. Estimated glomerular filtration rate (eGFR) ≤ 60 mL/min as calculated by the CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration) equation
15. Any clinically significant illness in the 28 days prior to study drug administration
16. Use of any prescription drugs (with the exception of hormonal contraceptives or hormone replacement therapy) in the 28 days prior to study drug administration, that in the opinion of an Investigator would put into question the status of the participant as healthy
17. Use of St. John's wort in the 28 days prior to study drug administration
18. Positive test result for alcohol and/or drugs of abuse at admission (prior to study drug administration). Subjects with positive results at admission may be rescheduled at the discretion of an Investigator. If tetrahydrocannabinol (THC) is positive at admission a cannabis intoxication evaluation will be done by an Investigator and subjects may be permitted to continue in the study at the discretion of an Investigator. Other positive test results should be reviewed to determine if the subject may be rescheduled, in the opinion of the investigator.
19. Positive screening results to HIV Ag/Ab combo, hepatitis B surface antigen or hepatitis C virus tests
20. Any other clinically significant abnormalities in laboratory test results at Screening that would, in the opinion of an Investigator, increase the subject's risk of participation, jeopardize complete participation in the study, or compromise interpretation of study data
21. Inclusion in a previous group for this clinical study
22. Intake of kratom in the 14 days prior to study drug administration
23. Intake of an Investigational Product (IP) in the 28 days prior to study drug administration
24. Donation of plasma in the 7 days prior to study drug administration
25. Donation of 1 unit of blood to American Red Cross or equivalent organization or donation of over 500 mL of blood in the 56 days prior to study drug administration
26. Subject cannot eat dairy and/or is lactose intolerant
27. Is, in the opinion of an Investigator or designee, considered unsuitable or unlikely to comply with the study protocol for any reason

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-08-16 (Actual); Primary Completion 2024-01-23 (Actual); Study Completion 2024-01-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Altasciences Clinical Kansas, Inc., Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort 1, 1 g of Kratom | Cohort 2, 3 g of Kratom | Cohort 3, 8 g of Kratom | Cohort 4, 10 g of Kratom | Cohort 5, 12 g of Kratom | Placebo
Started | 6 | 6 | 6 | 6 | 6 | 10
Completed | 6 | 6 | 6 | 6 | 6 | 10
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1, 1 g of Kratom | Cohort 2, 3 g of Kratom | Cohort 3, 8 g of Kratom | Cohort 4, 10 g of Kratom | Cohort 5, 12 g of Kratom | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 10 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.5 (8.78) | 32.2 (3.54) | 37.7 (10.69) | 40.3 (6.89) | 40.2 (6.40) | 32.5 (4.81) | 36.3 (7.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 1 | 1 | 0 | 3 | 5
  Male | 6 | 6 | 5 | 5 | 6 | 7 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 6 | 6 | 6 | 6 | 5 | 10 | 39
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 4 | 5 | 4 | 6 | 4 | 8 | 31
  White | 1 | 1 | 2 | 0 | 1 | 2 | 7
  Multiple | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Other | 0 | 0 | 0 | 0 | 1 | 0 | 1
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 24.02 (4.279) | 26.82 (4.222) | 27.42 (4.901) | 25.85 (2.811) | 24.33 (2.277) | 25.48 (4.132) | 25.64 (3.835)
Weight (kg) [Mean (Standard Deviation); unit: kg] | 73.78 (14.910) | 84.83 (14.552) | 79.60 (13.565) | 80.08 (12.090) | 74.62 (9.338) | 74.51 (12.946) | 77.56 (12.787)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: For purposes of monitoring safety, treatment-emergent adverse events (AEs) will be graded using the National Cancer Institute's Common Terminology Criteria for Adverse Events (version 5.0).
Time Frame: Day 1 through Day 7
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1, 1 g of Kratom | Cohort 2, 3 g of Kratom | Cohort 3, 8 g of Kratom | Cohort 4, 10 g of Kratom | Cohort 5, 12 g of Kratom | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 10
Participants | 1 | 1 | 5 | 4 | 3 | 4

2. Secondary Outcome: Maximum Observed Concentration
Description: Cmax (ng/mL) will be evaluated for: mitragynine, 7 hydroxy-mitragynine, paynantheine, speciogynine, and speciociliatine
Time Frame: 0, 0.25, 0.50, 1.00, 1.50, 2.00, 2.50, 3.00, 4.00, 6.00, 8.00, 10.00, 12.00, 24.00 and 48.00 hours post-dose
Population: Placebo subjects were not included in the PK population.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1, 1 g of Kratom | Cohort 2, 3 g of Kratom | Cohort 3, 8 g of Kratom | Cohort 4, 10 g of Kratom | Cohort 5, 12 g of Kratom | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 0
ng/mL
  Mitragynine | 41.664 (14.766) | 118.002 (46.816) | 197.496 (88.333) | 318.112 (163.400) | 378.507 (184.981) |
  7 hydroxy-mitragynine | 6.728 (2.182) | 17.751 (8.687) | 33.985 (11.184) | 48.388 (19.989) | 58.400 (22.717) |
  Paynantheine | 7.7 (2.6) | 19.0 (5.0) | 29.7 (14.6) | 66.7 (36.6) | 65.8 (34.2) |
  Speciogynine | 6.3 (1.9) | 15.8 (4.3) | 23.2 (10.1) | 58.9 (35.5) | 55.5 (31.0) |
  Speciociliatine | 39.1 (11.7) | 106.6 (23.9) | 168.9 (68.1) | 388.1 (217.2) | 409.7 (193.8) |
Statistical Analysis 1: Comparison: Cohort 1, 1 g of Kratom vs Cohort 2, 3 g of Kratom vs Cohort 3, 8 g of Kratom vs Cohort 4, 10 g of Kratom vs Cohort 5, 12 g of Kratom; Statistical Analysis for Dose-Proportionality of Mitragynine Pharmacokinetic Parameters (Pharmacokinetic Population); Test type: Other — Proportionality analysis was done using a power model; Slope = 0.829, 90% CI 2-sided [0.659 to 0.998]
Statistical Analysis 2: Comparison: Cohort 1, 1 g of Kratom vs Cohort 2, 3 g of Kratom vs Cohort 3, 8 g of Kratom vs Cohort 4, 10 g of Kratom vs Cohort 5, 12 g of Kratom; Statistical Analysis for Dose-Proportionality of 7-Hydroxy-Mitragynine Pharmacokinetic Parameters (Pharmacokinetic Population); Test type: Other — Proportionality analysis was done using a power model; Slope = 0.843, 90% CI 2-sided [0.713 to 0.973]
Statistical Analysis 3: Comparison: Cohort 1, 1 g of Kratom vs Cohort 2, 3 g of Kratom vs Cohort 3, 8 g of Kratom vs Cohort 4, 10 g of Kratom vs Cohort 5, 12 g of Kratom; Statistical Analysis for Dose-Proportionality of Paynantheine Pharmacokinetic Parameters (Pharmacokinetic Population); Test type: Other — Proportionality analysis was done using a power model; Slope = 0.811, 90% CI 2-sided [0.637 to 0.984]
Statistical Analysis 4: Comparison: Cohort 1, 1 g of Kratom vs Cohort 2, 3 g of Kratom vs Cohort 3, 8 g of Kratom vs Cohort 4, 10 g of Kratom vs Cohort 5, 12 g of Kratom; Statistical Analysis for Dose-Proportionality of Speciogynine Pharmacokinetic Parameters (Pharmacokinetic Population); Test type: Other — Proportionality analysis was done using a power model; Slope = 0.814, 90% CI 2-sided [0.633 to 0.994]
Statistical Analysis 5: Comparison: Cohort 1, 1 g of Kratom vs Cohort 2, 3 g of Kratom vs Cohort 3, 8 g of Kratom vs Cohort 4, 10 g of Kratom vs Cohort 5, 12 g of Kratom; Statistical Analysis for Dose-Proportionality of Speciociliatine Dose Adjusted Pharmacokinetic Parameters (Pharmacokinetic Population); Test type: Other — Proportionality analysis was done using a power model; Slope = 0.880, 90% CI 2-sided [0.720 to 1.039]

3. Secondary Outcome: Time of Maximum Observed Concentration
Description: Tmax (hours) will be evaluated for: mitragynine, 7 hydroxy-mitragynine, paynantheine, speciogynine, and speciociliatine
Time Frame: 0, 0.25, 0.50, 1.00, 1.50, 2.00, 2.50, 3.00, 4.00, 6.00, 8.00, 10.00, 12.00, 24.00 and 48.00 hours post-dose
Population: Placebo subjects were not included in the PK population.
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1, 1 g of Kratom | Cohort 2, 3 g of Kratom | Cohort 3, 8 g of Kratom | Cohort 4, 10 g of Kratom | Cohort 5, 12 g of Kratom | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 0
hours
  mitragynine | 4.02 [2.50 to 6.18] | 2.99 [2.50 to 4.00] | 5.04 [2.50 to 6.14] | 3.50 [2.50 to 4.00] | 2.00 [1.00 to 6.01] |
  7 hydroxy-mitragynine | 4.02 [2.50 to 6.18] | 3.50 [2.99 to 4.00] | 6.01 [3.00 to 10.02] | 4.00 [3.00 to 4.00] | 2.75 [1.50 to 6.01] |
  paynantheine | 4.02 [2.50 to 6.18] | 2.99 [2.50 to 4.00] | 5.04 [3.00 to 6.14] | 3.00 [2.50 to 4.00] | 3.29 [1.50 to 6.01] |
  speciogynine | 4.02 [2.50 to 6.18] | 3.00 [2.99 to 4.00] | 5.04 [3.00 to 10.02] | 4.00 [3.00 to 6.00] | 2.54 [1.50 to 6.01] |
  speciociliatine | 4.02 [3.00 to 8.04] | 5.00 [3.00 to 9.99] | 8.07 [3.00 to 12.00] | 5.00 [4.00 to 8.00] | 5.06 [2.00 to 10.01] |

4. Secondary Outcome: Area Under the Concentration Time Curve From Time Zero to the Time of Last Quantifiable Concentration (AUC0-T)
Description: AUC0-T (ng*h/mL) will be evaluated for: mitragynine, 7 hydroxy-mitragynine, paynantheine, speciogynine, and speciociliatine
Time Frame: 0, 0.25, 0.50, 1.00, 1.50, 2.00, 2.50, 3.00, 4.00, 6.00, 8.00, 10.00, 12.00, 24.00 and 48.00 hours post-dose
Population: Placebo subjects were not included in the PK population.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Cohort 1, 1 g of Kratom | Cohort 2, 3 g of Kratom | Cohort 3, 8 g of Kratom | Cohort 4, 10 g of Kratom | Cohort 5, 12 g of Kratom | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 0
ng*h/mL
  mitragynine | 305.383 (115.616) | 784.794 (380.290) | 1942.205 (737.483) | 3254.385 (2213.450) | 3271.209 (1577.443) |
  7 hydroxy-mitragynine | 53.518 (21.615) | 132.994 (85.838) | 412.602 (153.549) | 459.109 (226.314) | 574.260 (194.789) |
  paynantheine | 47.0 (19.0) | 132.9 (44.0) | 320.2 (134.0) | 725.2 (452.4) | 727.6 (397.9) |
  speciogynine | 53.4 (19.2) | 154.0 (44.1) | 341.0 (147.5) | 819.2 (521.6) | 790.0 (453.2) |
  speciociliatine | 573.9 (285.4) | 1910.9 (475.4) | 3359.2 (1257.7) | 7904.8 (4790.9) | 7449.8 (3695.4) |
Statistical Analysis 1: Comparison: Cohort 1, 1 g of Kratom vs Cohort 2, 3 g of Kratom vs Cohort 3, 8 g of Kratom vs Cohort 4, 10 g of Kratom vs Cohort 5, 12 g of Kratom; Statistical Analysis for Dose-Proportionality of Mitragynine Pharmacokinetic Parameters (Pharmacokinetic Population); Test type: Other — Proportionality analysis was done using a power model; Slope = 0.946, 90% CI 2-sided [0.768 to 1.123]
Statistical Analysis 2: Comparison: Cohort 1, 1 g of Kratom vs Cohort 2, 3 g of Kratom vs Cohort 3, 8 g of Kratom vs Cohort 4, 10 g of Kratom vs Cohort 5, 12 g of Kratom; [analysis description as in outcome 2, analysis 2]; Test type: Other — Proportionality analysis was done using a power model; Slope = 0.978, 90% CI 2-sided [0.821 to 1.134]
Statistical Analysis 3: Comparison: Cohort 1, 1 g of Kratom vs Cohort 2, 3 g of Kratom vs Cohort 3, 8 g of Kratom vs Cohort 4, 10 g of Kratom vs Cohort 5, 12 g of Kratom; Statistical Analysis for Dose-Proportionality of Paynantheine Pharmacokinetic Parameters (Pharmacokinetic Population); Test type: Other — Proportionality analysis was done using a power model; Slope = 1.075, 90% CI 2-sided [0.901 to 1.249]
Statistical Analysis 4: Comparison: Cohort 1, 1 g of Kratom vs Cohort 2, 3 g of Kratom vs Cohort 3, 8 g of Kratom vs Cohort 4, 10 g of Kratom vs Cohort 5, 12 g of Kratom; Statistical Analysis for Dose-Proportionality of Speciogynine Pharmacokinetic Parameters (Pharmacokinetic Population); Test type: Other — Proportionality analysis was done using a power model; Slope = 1.046, 90% CI 2-sided [0.870 to 1.222]
Statistical Analysis 5: Comparison: Cohort 1, 1 g of Kratom vs Cohort 2, 3 g of Kratom vs Cohort 3, 8 g of Kratom vs Cohort 4, 10 g of Kratom vs Cohort 5, 12 g of Kratom; [analysis description as in outcome 2, analysis 5]; Test type: Other — Proportionality analysis was done using a power model; Slope = 1.011, 90% CI 2-sided [0.844 to 1.178]

5. Secondary Outcome: Area Under the Concentration Time Curve Extrapolated to Infinity
Description: AUC0-inf (ng*h/mL) will be evaluated for: mitragynine, 7 hydroxy-mitragynine, paynantheine, speciogynine, and speciociliatine
Time Frame: 0, 0.25, 0.50, 1.00, 1.50, 2.00, 2.50, 3.00, 4.00, 6.00, 8.00, 10.00, 12.00, 24.00 and 48.00 hours post-dose
Population: Placebo subjects were not included in the PK population.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Cohort 1, 1 g of Kratom | Cohort 2, 3 g of Kratom | Cohort 3, 8 g of Kratom | Cohort 4, 10 g of Kratom | Cohort 5, 12 g of Kratom | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 0
ng*h/mL
  mitragynine | 341.941 (131.703) | 897.401 (436.438) | 2305.048 (1068.794) | 3950.438 (2839.536) | 3674.606 (1790.980) |
  7 hydroxy-mitragynine | 57.023 (21.974) | 139.322 (88.492) | 438.569 (169.329) | 515.160 (284.275) | 596.489 (206.138) |
  paynantheine | 58.3 (22.6) | 160.1 (52.6) | 380.3 (161.2) | 819.4 (477.5) | 814.8 (462.9) |
  speciogynine | 76.1 (27.5) | 190.1 (51.1) | 413.2 (189.8) | 958.6 (570.7) | 906.3 (544.4) |
  speciociliatine | 654.9 (377.1) | 2099.8 (578.7) | 4187.3 (1567.2) | 8908.0 (5130.1) | 8012.7 (4075.7) |
Statistical Analysis 1: Comparison: Cohort 1, 1 g of Kratom vs Cohort 2, 3 g of Kratom vs Cohort 3, 8 g of Kratom vs Cohort 4, 10 g of Kratom vs Cohort 5, 12 g of Kratom; Statistical Analysis for Dose-Proportionality of Mitragynine Pharmacokinetic Parameters (Pharmacokinetic Population); Test type: Other — Proportionality analysis was done using a power model; Slope = 0.959, 90% CI 2-sided [0.775 to 1.143]
Statistical Analysis 2: Comparison: Cohort 1, 1 g of Kratom vs Cohort 2, 3 g of Kratom vs Cohort 3, 8 g of Kratom vs Cohort 4, 10 g of Kratom vs Cohort 5, 12 g of Kratom; [analysis description as in outcome 2, analysis 2]; Test type: Other — Proportionality analysis was done using a power model; Slope = 0.974, 90% CI 2-sided [0.815 to 1.134]
Statistical Analysis 3: Comparison: Cohort 1, 1 g of Kratom vs Cohort 2, 3 g of Kratom vs Cohort 3, 8 g of Kratom vs Cohort 4, 10 g of Kratom vs Cohort 5, 12 g of Kratom; Statistical Analysis for Dose-Proportionality of Paynantheine Pharmacokinetic Parameters (Pharmacokinetic Population); Test type: Other — Proportionality analysis was done using a power model; Slope = 1.036, 90% CI 2-sided [0.866 to 1.207]
Statistical Analysis 4: Comparison: Cohort 1, 1 g of Kratom vs Cohort 2, 3 g of Kratom vs Cohort 3, 8 g of Kratom vs Cohort 4, 10 g of Kratom vs Cohort 5, 12 g of Kratom; Statistical Analysis for Dose-Proportionality of Speciogynine Pharmacokinetic Parameters (Pharmacokinetic Population); Test type: Other — Proportionality analysis was done using a power model; Slope = 0.967, 90% CI 2-sided [0.790 to 1.145]
Statistical Analysis 5: Comparison: Cohort 1, 1 g of Kratom vs Cohort 2, 3 g of Kratom vs Cohort 3, 8 g of Kratom vs Cohort 4, 10 g of Kratom vs Cohort 5, 12 g of Kratom; [analysis description as in outcome 2, analysis 5]; Test type: Other — Proportionality analysis was done using a power model; Slope = 1.025, 90% CI 2-sided [0.859 to 1.191]

6. Secondary Outcome: Dose-normalized Cmax Calculated at Cmax / Dose
Description: Cmax/D (ng/mL/g) will be evaluated for: mitragynine, 7 hydroxy-mitragynine, paynantheine, speciogynine, and speciociliatine
Time Frame: 0, 0.25, 0.50, 1.00, 1.50, 2.00, 2.50, 3.00, 4.00, 6.00, 8.00, 10.00, 12.00, 24.00 and 48.00 hours post-dose
Population: Placebo subjects were not included in the PK population.
Measure: Mean (Standard Deviation); unit: ng/mL/g
Arm/Group | Cohort 1, 1 g of Kratom | Cohort 2, 3 g of Kratom | Cohort 3, 8 g of Kratom | Cohort 4, 10 g of Kratom | Cohort 5, 12 g of Kratom | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 0
ng/mL/g
  mitragynine | 41.664 (14.766) | 39.334 (15.605) | 24.687 (11.042) | 31.811 (16.340) | 31.542 (15.415) |
  7 hydroxy-mitragynine | 6.728 (2.182) | 5.917 (2.896) | 4.248 (1.398) | 4.839 (1.999) | 4.867 (1.893) |
  paynantheine | 7.7 (2.6) | 6.3 (1.7) | 3.7 (1.8) | 6.7 (3.7) | 5.5 (2.8) |
  speciogynine | 6.3 (1.9) | 5.2 (1.4) | 2.9 (1.3) | 5.9 (3.5) | 4.6 (2.6) |
  speciociliatine | 39.1 (11.7) | 35.5 (8.0) | 21.1 (8.5) | 38.8 (21.7) | 34.1 (16.2) |

7. Secondary Outcome: Dose-normalized AUC0-T Calculated as AUC0-T / Dose
Description: AUC0-T/D (ng*h/mL/g) will be evaluated for: mitragynine, 7 hydroxy-mitragynine, paynantheine, speciogynine, and speciociliatine
Time Frame: 0, 0.25, 0.50, 1.00, 1.50, 2.00, 2.50, 3.00, 4.00, 6.00, 8.00, 10.00, 12.00, 24.00 and 48.00 hours post-dose
Population: Placebo subjects were not included in the PK population.
Measure: Mean (Standard Deviation); unit: ng*h/mL/g
Arm/Group | Cohort 1, 1 g of Kratom | Cohort 2, 3 g of Kratom | Cohort 3, 8 g of Kratom | Cohort 4, 10 g of Kratom | Cohort 5, 12 g of Kratom | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 0
ng*h/mL/g
  mitragynine | 305.383 (115.616) | 261.598 (126.763) | 242.776 (92.185) | 325.438 (221.345) | 272.601 (131.454) |
  7 hydroxy-mitragynine | 53.518 (21.615) | 44.331 (28.613) | 51.575 (19.194) | 45.911 (22.631) | 47.855 (16.232) |
  paynantheine | 47.0 (19.0) | 44.3 (14.7) | 40.0 (16.8) | 72.5 (45.2) | 60.6 (33.2) |
  speciogynine | 53.4 (19.2) | 51.3 (14.7) | 42.6 (18.4) | 81.9 (52.2) | 65.8 (37.8) |
  speciociliatine | 573.9 (285.4) | 637.0 (158.5) | 419.9 (157.2) | 790.5 (479.1) | 620.8 (308.0) |

8. Secondary Outcome: Dose-normalized AUC0-inf Calculated as AUC0-inf / Dose
Description: AUC0-inf/D (ng*h/mL/g) will be evaluated for: mitragynine, 7 hydroxy-mitragynine, paynantheine, speciogynine, and speciociliatine
Time Frame: 0, 0.25, 0.50, 1.00, 1.50, 2.00, 2.50, 3.00, 4.00, 6.00, 8.00, 10.00, 12.00, 24.00 and 48.00 hours post-dose
Population: Placebo subjects were not included in the PK population.
Measure: Mean (Standard Deviation); unit: (ng*h/mL/g
Arm/Group | Cohort 1, 1 g of Kratom | Cohort 2, 3 g of Kratom | Cohort 3, 8 g of Kratom | Cohort 4, 10 g of Kratom | Cohort 5, 12 g of Kratom | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 0
(ng*h/mL/g
  mitragynine | 341.941 (131.703) | 299.134 (145.479) | 288.131 (133.599) | 395.044 (283.954) | 306.217 (149.248) |
  7 hydroxy-mitragynine | 57.023 (21.974) | 46.441 (29.497) | 54.821 (21.166) | 51.516 (28.427) | 49.707 (17.178) |
  paynantheine | 58.3 (22.6) | 53.4 (17.5) | 47.5 (20.2) | 81.9 (47.8) | 67.9 (38.6) |
  speciogynine | 76.1 (27.5) | 63.4 (17.0) | 51.6 (23.7) | 95.9 (57.1) | 75.5 (45.4) |
  speciociliatine | 654.9 (377.1) | 699.9 (192.9) | 523.4 (195.9) | 890.8 (513.0) | 667.7 (339.6) |

9. Secondary Outcome: Maximum Effect for Drug Liking
Description: Maximum (peak) effect (Emax) for Drug Liking assessed on a bipolar (0 to 100 points) visual analog scale (VAS). Anchors will be presented using text such as "strong disliking" (score = 0), "neither like nor dislike" (score = 50) to "strong liking" (score = 100).
Time Frame: 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, and 24 hours postdose
Measure: Mean (Standard Error); unit: score on a scale (VAS Emax)
Arm/Group | Cohort 1, 1 g of Kratom | Cohort 2, 3 g of Kratom | Cohort 3, 8 g of Kratom | Cohort 4, 10 g of Kratom | Cohort 5, 12 g of Kratom | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 10
score on a scale (VAS Emax) | 50.7 (0.67) | 51.7 (1.67) | 60.2 (8.17) | 52.2 (0.98) | 68.7 (9.22) | 50.2 (0.13)
Statistical Analysis 1: Comparison: Cohort 5, 12 g of Kratom vs Placebo; Test type: Superiority; Least-Square Mean = 18.5, 95% CI 2-sided [6.16 to 30.78], Standard Error of Mean 6.06

10. Secondary Outcome: Maximum Effect for Overall Drug Liking
Description: Maximum (peak) effect (Emax) for Overall Drug Liking assessed on a bipolar (0 to 100 points) visual analog scale (VAS). Anchors will be presented using text such as "strong disliking" (score = 0), "neither like nor dislike" (score = 50) to "strong liking" (score = 100).
Time Frame: 12 and 24 hours postdose
Measure: Mean (Standard Error); unit: score on a scale (VAS EMax)
Arm/Group | Cohort 1, 1 g of Kratom | Cohort 2, 3 g of Kratom | Cohort 3, 8 g of Kratom | Cohort 4, 10 g of Kratom | Cohort 5, 12 g of Kratom | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 10
score on a scale (VAS EMax) | 50.2 (0.17) | 50 (0) | 61.8 (8.37) | 55.7 (13.22) | 67 (7.96) | 45.1 (4.9)

11. Secondary Outcome: Maximum Effect for Take Drug Again
Description: Maximum (peak) effect (Emax) for Take Drug Again assessed on a bipolar (0 to 100 points) visual analog scale (VAS). Anchors will be presented using text such as "definitely would not" (score = 0), "neither would nor would not" (score = 50) to "definitely would" (score = 100).
Time Frame: 12 and 24 hours postdose
Measure: Mean (Standard Error); unit: score on a scale (VAS EMax)
Arm/Group | Cohort 1, 1 g of Kratom | Cohort 2, 3 g of Kratom | Cohort 3, 8 g of Kratom | Cohort 4, 10 g of Kratom | Cohort 5, 12 g of Kratom | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 10
score on a scale (VAS EMax) | 53.3 (3.14) | 50.0 (0) | 65.2 (8.04) | 49.8 (17.17) | 61 (8.57) | 45.9 (5.2)

12. Secondary Outcome: Maximum Effect for High
Description: Maximum (peak) effect (Emax) for High assessed on an unipolar (0 to 100 points) visual analog scale (VAS). Anchors will be presented using text such as "not at all" (score = 0) to "extremely" (score = 100).
Time Frame: Predose and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, and 24 hours postdose
Measure: Mean (Standard Error); unit: score on a scale (VAS EMax)
Arm/Group | Cohort 1, 1 g of Kratom | Cohort 2, 3 g of Kratom | Cohort 3, 8 g of Kratom | Cohort 4, 10 g of Kratom | Cohort 5, 12 g of Kratom | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 10
score on a scale (VAS EMax) | 0.5 (0.5) | 1.2 (1.17) | 10.8 (4.94) | 8.5 (5.33) | 46.3 (14.14) | 0.4 (0.31)
Statistical Analysis 1: Comparison: Cohort 5, 12 g of Kratom vs Placebo; Statistical Analysis for High Visual Analog Scale (Emax); Test type: Superiority; p < 0.001, ANOVA; Least-Squared Mean = 45.9, 95% CI 2-sided [30.20 to 61.67], Standard Error of Mean 7.74

ADVERSE EVENTS:
Time Frame: 37 days.
Description: For the purposes of this study, the monitoring period for AEs extends from the pre-trial evaluation until collection of the last blood sample of the study. From screening to dosing of the study, AEs will be recorded as screening events or as part of the medical history, as applicable.
Arm/Group | Cohort 1, 1 g of Kratom | Cohort 2, 3 g of Kratom | Cohort 3, 8 g of Kratom | Cohort 4, 10 g of Kratom | Cohort 5, 12 g of Kratom | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/10
Other Adverse Events (participants affected / at risk) | 1/6 | 1/6 | 5/6 | 5/6 | 3/6 | 4/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1, 1 g of Kratom (N=6) | Cohort 2, 3 g of Kratom (N=6) | Cohort 3, 8 g of Kratom (N=6) | Cohort 4, 10 g of Kratom (N=6) | Cohort 5, 12 g of Kratom (N=6) | Placebo (N=10)
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 — Right arm paresthesia.
Blood pressure systolic increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 — Elevated systolic blood pressure.
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 — Pruritus right hand.
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 3 | 0 | 2 — Drowsiness / Feeling sleepy
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 2 | 0 — Emesis
Leukocyturia (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Euphoric mood (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 0 — Feeling high.
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 1
Irritability (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 — Feeling of anxiety.
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 — Diaphoresis
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (4):
  • Study Protocol (2023-06-05): https://cdn.clinicaltrials.gov/large-docs/70/NCT06072170/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-04): https://cdn.clinicaltrials.gov/large-docs/70/NCT06072170/SAP_001.pdf
  • Informed Consent Form: Pregnancy Partner Information Form (2023-06-07): https://cdn.clinicaltrials.gov/large-docs/70/NCT06072170/ICF_002.pdf
  • Informed Consent Form: Informed Consent Form (2023-06-07): https://cdn.clinicaltrials.gov/large-docs/70/NCT06072170/ICF_003.pdf